CLINICAL TRIAL: NCT06108999
Title: Prospective, Multicentric, Post-market Clinical Investigation to Evaluate the Performance and Safety of Connettivina Bio Line in Management of Acute and Chronic Wounds
Brief Title: Management of Acute and Chronic Wounds With Hyaluronic Acid
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AQ04-20-01
Record Dates: First submitted 2023-10-16; First posted 2023-10-31 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Wound Heal; Wound; Foot
MeSH Terms: conditions — Foot Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connettivia BIO Cream (Experimental): All subjects will be treated with Connettivina BIO line (Cream or Gauze)
  Interventions: Device: Connettivina BIO cream and gauze
- Connettivina BIO Gauze (Experimental): All subjects will be treated with Connettivina BIO line (Cream or Gauze)
  Interventions: Device: Connettivina BIO cream and gauze

INTERVENTIONS:
Device: Connettivina BIO cream and gauze — Connettivina Bio cream and gauze-pad efficacy and tolerability will be evaluated in the management of acute or chronic wounds of different etiology, according to instruction for use. Only one wound per patient will be considered for the treatment according to the study protocol. The schedule treatment will consist on a daily medication changes, according to the instruction for use and the clinical practice, for a maximum of 7 Visits.

SUMMARY:
The purpose of this study is to evaluate the performance and safety of Connettivina Bio, when used in the management of wounds. Moreover, the study will evaluate the correlation of the 'dressing system' (formed by the Connettivina Bio primary dressing plus a secondary one) used in different care settings. The study will include Italian healthcare facilities.

DETAILED DESCRIPTION:
The primary objective of the prospective, multicentric, post-market clinical investigation is to evaluate the performance of Connettivina Bio (cream, gauze-pads) in the amelioration of wound bed appearance after 14 days of treatment. This objective will be assessed by measuring the percentage of patients showing, from baseline to 14 days of treatment, positive change in at least one of the following parameters: amelioration of wound tissue type (4=necrotic, 3=slough, 2=granulation tissue, 1=epithelial tissue, 0=closed), decrease of exudate amount (1=dry, 2=moist,3= slightly exuding, 4=heavily exuding, 5=wet) and amelioration of exudate type (1=bloody, 2=bloody/purulent, 3=clear, 4=murky,5= purulent, 6=serous). Furthermore, the secondary objectives of this clinical investigation include to define the Investigator's choice in clinical practice of Connettivina Bio (cream, gauze-pad) related to the clinical wound characteristics, the type of secondary dressing applied on the wound and the wound etiology, for this reason a descriptive analysis will be performed at baseline. Additionally, for the secondary objectives, the performance of Connettivina Bio (cream, gauze-pads) will be evaluated from baseline to 7, 21, 28, 42 and 56 days as amelioration of wound bed appearance in terms of type of wound bed tissue and exudate quantity and quality. To evaluate the improvement of quality of life of patients treated, the latter will be evaluated as a change from baseline to 56 days after the start of treatment, through administration of EuroQoL-5D (EQ-5D). Moreover, to evaluate the easiness of Connettivina Bio (cream, gauze-pads) application, the latter will be appraised by the clinician and by the patient after 56 days from the start of treatment as excellent, good, acceptable, bad or unacceptable. Finally, the safety and tolerability of Connettivina Bio (cream, gauze-pads) will be assessed throughout all the visits by investigating local and expected adverse events, as consequence of the product application and any other adverse event occurred during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Male or female ≥18 years.
3. Patients selected to be treated with Connettivina Bio.
4. Patients with wound of the following etiology: first and second degree burns; surgical wounds; vascular ulcers; metabolic ulcers; pressure ulcers.
5. Patients followed on an outpatient or home basis.
6. Wound area ≥ 10 cm2 and ≤ 100 cm2

Exclusion Criteria:

1. Patients < 18 years.
2. Patients with acute or chronic infected lesions.
3. Hospitalized patients.
4. Patients with acute or chronic lesions at high risk of infection, presenting at least one of the following criteria:

   * Stalled wound, without any clinical sign of healing progression
   * Immune system disorders
   * Protein-energy malnutrition
   * Alcohol, smoking and drug abuse
   * Conditions associated with hypoxia and/or poor tissue perfusion
   * Corticosteroid, cytotoxic or immunosuppressive therapy.
5. Subjects unable to understand informed consent or having a high probability of non-compliance with the study procedures and or non-completion of the study according to investigator's judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2022-07-29 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the performance of Connettivina Bio line in the amelioration of wound bed appearance | 14 days
  The performance of Connettivina Bio line, in the amelioration of wound bed appearance, will be evaluated from baseline up to 14 days of treatment. The percentage of patients showing a change in at least of one of the following evaluated parameters: amelioration of wound tissue type (necrotic, slough, granulation tissue, epithelial tissue, closed), decrease of exudate amount (dry, moist, slightly exuding, heavily exuding, wet) and amelioration of exudate type (bloody, bloody/purulent, clear, murky, purulent, serous).

SECONDARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events | 8 weeks
  The safety and tolerability of Connettivina Bio will be assessed throughout all the visits by investigating local and expected adverse events, as a consequence of the product application. Additionally, any other adverse event occurred during the study will be considered and evaluated

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Centro Grandi Ustionati OSPEDALE BUFALINI DI CESENA - (FC), Cesena, Forlì-Cesena
  - AOU Ospedali Riuniti SOD-Clinica di Chirurgia Plastica e Ricostruttiva, Ancona
  - Azienda Sanitaria Universitaria Giuliano Isontina (ASU GI) - SC (UCO), Trieste